CLINICAL TRIAL: NCT01729260
Title: Phase I Study of Mebendazole in Newly Diagnosed High-Grade Glioma Patients Receiving Temozolomide
Brief Title: Mebendazole in Newly Diagnosed High-Grade Glioma Patients Receiving Temozolomide
Acronym: Mebendazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Accelerate Brain Cancer Cure (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1194; NA_00049848 (Other: JHMIRB)
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Newly Diagnosed High-Grade Glioma
Keywords: Glioblastoma; mebendazole; temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Mebendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mebendazole (Experimental): All study participants will receive study drug; Mebendazole.
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Mebendazole — The mebendazole will be given by mouth three times every day on a 28 day cycle. it's in the form of 500 mg chewable tablets, to be taken with meals.
  Other Names: Brand name: Vermox

SUMMARY:
The purpose of this study is to find the highest dose of mebendazole (MBZ) that can be safely given to people with malignant brain tumors in combination with the current standard of care (temozolomide) without causing severe side effects. We also want to find out if MBZ can slow the growth of the brain tumor. The study doctors have found that MBZ is effective against malignant brain tumors in the laboratory and animal models of brain tumors.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common and aggressive brain cancer, and despite significant advances in treatment the majority of patients die within two years of diagnosis. During routine animal studies we serendipitously observed that fenbendazole, a benzimidazole antihelminthic used for pinworms, prevented tumor engraftment. Subsequent in vitro and in vivo experiments with benzimidazoles identified mebendazole as the drug having the best results in preclinical testing 1. In GBM cell lines, mebendazole displayed cytotoxicity with IC50s ranging from 0.1-0.3 μM. Mebendazole disrupted microtubule formation in GBM cells and it's in vitro activity was correlated with reduced tubulin polymerization. In two orthotopic mouse glioma models, one syngeneic and one xenograft, mebendazole significantly extended average survival up to 63% compared to untreated controls 1.

Mebendazole is an FDA approved antiparasitic agent with a well-established side effect and safety record and was effective in our animal models in dosing schedules that are documented as safe in humans. Therefore, mebendazole is a possible anti-cancer therapeutic with pre-clinical safety and efficacy and provides a promising opportunity for a clinical trial in patients with malignant gliomas.

In addition, a recently published case report case report from the University of Michigan documented successful long term control in metastatic adrenocortical adenocarcinoma using mebendazole 2. Mebendazole was well tolerated at 200 mg/day and used as the sole treatment after the patient failed other chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed newly diagnosed high-grade glioma(WHO Grade III or IV)
2. Age ≥18 years
3. Karnofsky Performance Score (KPS) ≥ 60%
4. Life expectancy greater than 12 weeks
5. Patients must have adequate organ and marrow function
6. Completed >80% of the prescribed radiation therapy and concurrent temozolomide according to the Stupp regimen without grade 3 or 4 hematologic toxicity
7. Patients may have received Gliadel during surgery
8. Ability to swallow pills and keep medication record
9. women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation.
10. Ability to understand and willingness to sign a written informed consent document
11. Be able to comply with treatment plan, study procedures and follow-up examinations

Exclusion Criteria:

1. Patients must not have received prior therapy other than standard chemoradiation according to Stupp et al and Gliadel.
2. Patients may not be receiving any other investigational agents while on study
3. Patients who have known allergy to mebendazole or benzimidazole
4. Patients who have previously had a severe side effect, such as agranulocytosis and neutropenia, in conjunction with previous mebendazole or benzimidazole class drug for a parasitic infection
5. Patients who are taking metronidazole and cannot be safely moved to a different antibiotic greater than 7 days prior to starting mebendazole therapy
6. Patients who have taken any benzimidazole (ABZ, flubendazole, thiabendazole, fenbendazole, triclabendazole, etc.) within the last 3 months
7. Patients who are taking any anti-convulsant medication that interferes with the cytochrome P450 pathway (e.g. phenytoin, phenobarbital, carbamazepine, etc.)
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, chronic hepatitis, acute hepatitis, or psychiatric illness/social situation that would limit compliance with study requirements
9. Pregnant women are excluded
10. Patients with human immunodeficiency virus (HIV), hepatitis B surface antigen or hepatitis C positive; or with a history of chronic active hepatitis or cirrhosis
11. Patients with a history of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product administration or may interfere with the interpretation of the results
12. Patients who are not available for follow-up assessments or unable to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of mebendazole | 8 months
  To determine the maximum tolerated dose (MTD) of mebendazole in combination with temozolomide (TMZ) given after surgery and the standard radiation and TMZ treatment in patients with newly diagnosed malignant gliomas.

SECONDARY OUTCOMES:
Overall Survival | 10 years
  Overall survival in years.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gallia, MD, Principal Investigator — Johns Hopkins University School of Medicine, Department of Neurosurgery
Locations (1):
- The Johs Hopkins Hospital, Baltimore, Maryland, United States